CLINICAL TRIAL: NCT00897364
Title: Analysis of Intermediate Endpoint Biomarkers in the Respiratory Epithelium of Smokers Compared to Non-Smoking Controls
Brief Title: Biomarkers in the Nose, Throat, and Lung Tissue of Smokers and Non-Smokers
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 95-413; P50CA058187 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: non-small cell lung cancer; small cell lung cancer; squamous lung dysplasia
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endobronchial biopsies, blood, sputum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RATIONALE: Studying samples of tissue from smokers and non-smokers in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This phase II study is looking at biomarkers in the nose, throat, and lung tissue of smokers and non-smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Define the molecular and biochemical profiles of airway epithelium of smokers with no disease, smokers with airflow obstruction and abnormal sputum cytology, and non-smokers.

Secondary

* Assess the occurrence of abnormalities in non-smokers, smokers with no disease, smokers with various grades of dysplasia, and smokers with lung cancer.

OUTLINE: Patients are stratified according to smoking status (smoker vs non-smoker) and disease (no disease vs airflow obstruction and abnormal sputum cytology vs various grades of dysplasia vs lung cancer).

Biological samples are collected and analyzed for future research studies.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. - Adults > 45 years of age, to be age matched with a previously enrolled cohort of current and ex-smokers with airflow obstruction and moderate atypia on sputum cytology, to be included in the following groups.
2. - Non-smoking (less than 100 cigarettes per lifetime) controls >50 years of age, to be age matched with a previously enrolled cohort with airflow obstruction (FEV1 < 75% predicted and FEV1/FVC < 75%) and moderate atypia on sputum cytology.
3. - Current smokers with > 30 pack years, no airflow obstruction (FEV1 > 90% predicted) or lung cancer, >50 years of age, to be age matched with a previously enrolled cohort with airflow obstruction and moderate atypia on sputum cytology .
4. - No prior history of a head and neck or bronchogenic carcinoma.
5. - Patients must be fully informed of the investigational nature of this study and must sign an informed consent in accordance with institutional and FDA guidelines.

Exclusion Criteria:

1. - Clinically apparent bleeding diathesis.
2. - Cardiac dysrhythmia that is potentially life-threatening, such as ventricular tachycardia, multifocal premature ventricular contractions or supraventricular tachycardias with a rapid ventricular response. Well-controlled atrial fibrillation or rare (< 2/minute) premature ventricular contractions are not exclusionary.
3. - Hypoxemia (less than 90% saturation with supplemental oxygen) during bronchoscopy.
4. - Evidence of clinically active coronary artery disease, including myocardial infarction within 6 weeks, chest pain, or poorly controlled congestive heart failure, or any other serious medical condition which would preclude a patient from undergoing a bronchoscopy.
5. - Acute bronchitis or pneumonia within 8 weeks.
6. - Inability to give informed consent.
7. - Current smokers with no airflow obstruction may not have a history of coughing more than two times /week.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk for lung cancer and age matched normal volunters
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2000-05; Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

PRIMARY OUTCOMES:
Molecular and biochemical profiles | Upon completion of trial
  Evaluation of both Molecular and Biochemical profiles of normal non-smokers, smokers with no apparent disease (no airflow obstruction or cancer), and smokers with airflow obstruction and abnormal sputum cytology.

SECONDARY OUTCOMES:
Occurrence of abnormalities | Upon completion of trial
  Stratify abnormalities as to whether they occur frequently in normal non-smokers, smokers without disease, smokers with various grades of dysplasia, or smokers with lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: York E. Miller, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado, United States